CLINICAL TRIAL: NCT04745481
Title: Effectiveness Evaluation of Trunk Stabilization Training Using Balance Pro(SBT-330) for Stroke Patients With Reduced Balance Ability
Brief Title: Effects of Trunk Stabilization Training Device on Balance Ability for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Head of Rehabilitation Medicine, Principal Investigator, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-2020-010
Record Dates: First submitted 2021-01-31; First posted 2021-02-09 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: trunk stabilization training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk stabilization training device (Experimental): Participants will receive conventional rehabilitation and use trunk stabilization training device 30min each daily, 20 times for 4weeks.
  Interventions: Device: Trunk stabilization training device
- Conventional rehabilitation (Active Comparator): Participants will receive conventional rehabilitation 60min daily, 20times for 4weeks.
  Interventions: Device: Conventional rehabilitation

INTERVENTIONS:
Device: Trunk stabilization training device — Conventional rehabilitation 30min daily, 20times 4weeks
  +Trunk stabilization training device 30min daily, 20time 4weeks
  Other Names: Balance Pro(SBT-330)
  Arms: Trunk stabilization training device
Device: Conventional rehabilitation — Conventional rehabilitation 30min daily, 20times 4weeks
  +Conventional rehabilitation 30min daily, 20times 4weeks
  Other Names: Ergometer, Stepper
  Arms: Conventional rehabilitation

SUMMARY:
The purpose of this study is to assess the effectiveness of Balance pro(SBT-330:trunk stabilization training device) for stroke patients reduced balance ability

DETAILED DESCRIPTION:
after being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. Subjects who pass the screening test will randomize in a 1:1 ratio to experimental group(conventional rehabilitation + trunk stabilization training device, 30min each, 20days) or control group(conventional rehabilitation + conventional rehabilitation, 30min each, 20days). And then, They receive a registration number within 7 days and proceed with the pre-intervention test.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients 40 years or older (within 2 years of onset)
* Those who have no problems with visual function in conducting and conducting clinical trials
* Patients who are found to have decreased balance ability after stroke (BBS score is 21-40 points)
* Those who do not have orthopedic diseases in both lower limbs
* Subjects with cognitive functions capable of fulfilling and carrying out instructions
* Those who voluntarily consent to the clinical trial

Exclusion Criteria:

* Subjects with intellectual disabilities to the extent that they are unable to perform instructions
* Subjects taking drugs that may affect the study
* Subjects with skin and musculoskeletal abnormalities for which the device cannot be worn
* Patients with neurological disorders other than stroke and other disorders that may affect balance
* Other subjects who are judged to be unsuitable for this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Berg Balance Scale | Change from baseline Berg Balance Scale at week 4
  The Berg Balance Scale(BBS) is the quantified cutoff values for the four basic gait-related activities of stroke patients. It consists of a total of 14 items, and each item is divided into 5 levels, ranging from 0 to 4 points, with a total score of 56 points. Interpretation of exercise state according to score is 0-20: Wheelchair bound. 21-40: Walking with assistance. 41-56: independent.

SECONDARY OUTCOMES:
Timed Up and Go test | baseline and week 4
  The Timed Up and Go test(TUG) starts with sitting in a chair and measures the time it takes to get up and walk 3 meters back to sitting on the chair.
Functional Ambulation Category | baseline and week 4
  The Functional Ambulation Category(FAC) is a 7-point scale to evaluate the gait and mobility of patients with nervous and musculoskeletal injury. A higher score is interpreted as having higher independence of walking, and a score of 3 or less is considered difficult to move independently. It is a tool to evaluate not only balance ability but also actual mobility ability.
Korean version of Modified Barthel Index | baseline and week 4
  The Korean version of Modified Barthel Index(K-MBI) is a tool to evaluate the patient's level of independence in daily living activities, including basic daily living activities and instrumental daily living activities. It consists of 5 to 15 points depending on the item, and the perfect score is 100 points. The higher the score, the higher the patient's level of independence from daily activities is considered.
Fugl-Meyer Assessment(L/E) | baseline and week 4
  The Fugl-Meyer Assessment(FMA)(L/E) is an exercise ability scale to evaluate the motor function of stroke patients, and it is a tool to evaluate motor function of the healthy and injured upper and lower limbs. Each exercise item is evaluated on a 2-point scale and 3-point scale, with a perfect score of 100. In this study, lower limb evaluation items are implemented.
Trunk Impairment Scale | baseline and week 4
  The Trunk Impairment Scale(TIS) is for the motor impairment of the trunk of a stroke patient.
  As an optimal test method, it measures static and dynamic balance and coordination between the body in a sitting position. There are a total of 17 items with 3 items for static balance ability in a sitting position, 10 items for dynamic balance ability, and 4 items for trunk coordination, and minimum 0 to maximum 23 points.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-il Shin, PhD, Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan national university Yangsan Hospital, Gyeongsang, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Min JH, Seong HY, Ko SH, Jo WR, Sohn HJ, Ahn YH, Son JH, Seo HY, Son YR, Mun SJ, Ko MH, Shin YI. Effects of trunk stabilization training robot on postural control and gait in patients with chronic stroke: a randomized controlled trial. Int J Rehabil Res. 2020 Jun;43(2):159-166. doi: 10.1097/MRR.0000000000000399. PMID 32282572
- [Background] Chung SH, Kim JH, Yong SY, Lee YH, Park JM, Kim SH, Lee HC. Effect of Task-Specific Lower Extremity Training on Cognitive and Gait Function in Stroke Patients: A Prospective Randomized Controlled Trial. Ann Rehabil Med. 2019 Feb;43(1):1-10. doi: 10.5535/arm.2019.43.1.1. Epub 2019 Feb 28. PMID 30852865